CLINICAL TRIAL: NCT01990014
Title: Multicenter Clinical Study Evaluating the Functional Prognosis and Quality of Life at Least 2 Years in Patients Treated With Decompressive Craniectomy for Malignant Sylvian Ischemic Stroke
Brief Title: Craniectomy Protocol
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/08-I
Record Dates: First submitted 2013-10-25; First posted 2013-11-21 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke; Decompressive Craniectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- craniectomy: Adult subjects who experienced a cerebral infarction extended the sylvian area, and having received treatment by decompressive craniectomy.

SUMMARY:
The objective of this protocol is to evaluate the quality of life and functional disability in the long term (2 years after craniectomy) in subject's victims of malignant Sylvien stroke who received a decompressive craniotomy in the acute phase. Patients who have given their consent to be evaluated at least two years after their stroke and their operation in a single visit by clinical examination and procurement of standardized scales. Will be measured the quality of life through scale SIS3.0, residual disability by the Rankin scale. The quality of life of the carer will be assessed through scales and Zarit carer version of SIS3.0. The existence of predictive parameters of long-term evolution will be searched in determining the existence of a correlation between demographic data and baseline characteristics of the stroke on and the evolution of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years
* Having presented an ischemic stroke involving the sylvian area
* Having received decompressive craniectomy in acute ischemic stroke
* Time between stroke and the inclusion of at least 24 months
* Signed informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Patients with a Rankin score before stroke than or equal to 3
* Stroke in multiple territories (contralateral carotid and / or vertebrobasilar) associated with stroke in the acute phase describing which in the opinion of the investigator significantly influence the long-term functional prognosis
* Cognitive deterioration or severe aphasia making it impossible to fill out questionnaires
* Minors
* Major under curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who experienced a cerebral infarction extended the sylvian area, and having received treatment by decompressive craniectomy.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To assess the quality of life for long-term patients victims of malignant sylvian ischemic stroke who received decompressive craniectomy. | at least two years

SECONDARY OUTCOMES:
To evaluate the quality of life in the physical and psychosocial domains | at least two years
To evaluate the evolution of functional disability | At 3 months, 12 months and 24 months.
To evaluate the life satisfaction | at least two years
To assess the rate of recovery work | at least two years
To evaluate the retrospective review of patients achieving craniectomy | at least two years
To determine the prognostic factors that influence the level of handicap and quality of life in the long term. | at least two years
To evaluate the quality of life and level of long-term care accompanying persons caring for the near a victim of malignant sylvian ischemic stroke who received a decompressive craniotomy. | at least two years

CONTACTS AND LOCATIONS:
Overall Officials: SÉVIN ALLOUET Mathieu, Dr, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHU de Brest, Brest
  - CH R U Pontchaillou, Rennes
  - CHU Bretonneau, Tours